CLINICAL TRIAL: NCT05007743
Title: Randomized Trial of Effects of Transcutaneous Vagus Nerve Stimulation in Chronic Pain Patients and Healthy Controls
Brief Title: Effects of Transcutaneous Vagus Nerve Stimulation in Chronic Pain Patients and Healthy Controls
Acronym: tVNS-PP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Thomas Meyer, Head of Laboratory, University Medical Center Goettingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 27/7/18
Record Dates: First submitted 2021-07-15; First posted 2021-08-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Restless Legs Syndrome; Chronic Pain
Keywords: RLS, vagus nerve stimulation
MeSH Terms: conditions — Restless Legs Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: A crossover design is used for the investigation of the healthy cohort and a parallel design will be used for the patient group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation of inner tragus (Active Comparator): Comparing autonomic hemodynamic functions and immune responses pre- and post-stimulation of the vagus nerve
  Interventions: Device: Transcutaneous vagus nerve stimulation
- Stimulation of ear lobe (Sham Comparator): Comparing autonomic hemodynamic functions and immune responses pre- and post-stimulation of the vagus nerve
  Interventions: Device: Transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — Frequency of 30 Hz, biphasic, rectangular pulses with a pulse width of 250 µs and an intensity of 20 mA.
  Device: Easy Tens+ device (body clock, London, UK)

SUMMARY:
The tVNS-PP trial investigates the effects of transcutaneous vagus nerve stimulation (tVNS) on autonomic functions, immune responses, and disease severity in chronic pain and restless legs syndrome (RLS) patients as compared to healthy controls.

DETAILED DESCRIPTION:
A pilot study with healthy participants will investigate whether transcutaneous vagus nerve stimulation at the inner tragus reduces heart rate variability and lowers blood pressure without causing undesirable, severe side effects. In addition, changes in immune markers will be analyzed in blood samples before and after the interventions. Patients with primary restless legs syndrome will undergo a similar experimental protocol, except that transcutaneous vagus nerve stimulation will be performed daily. The aim is to determine whether stimulation reduces disease severity and chronic pain while improving quality of life.

ELIGIBILITY:
Inclusion criteria:

* Male and female participants between 18 and 80 years old
* Written informed consent

Exclusion criteria:

* Age younger than 18 years or older than 80 years
* Participants with somatic or mental comorbidities, especially malignant tumor diseases, cardiac insufficiencies > NYHA II, severe depressive episodes, psychosis or dementia
* Pregnancy or breast feeding
* Addictions to alcohol, medications or drugs (except tobacco)
* An existing legal guardianship
* Participation in another scientific study within the previous eight weeks before enrollment
* Restless Legs Syndrome patients with one of the following secondary predispositions: iron deficiency, polyneuropathy, prolapsed disk, spinal stenosis or chronic obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-21 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
International RLS Severity Scale | Seven days
  Numeric score quantifying disease severity. This numeric rating scale ranges from 0 to 40 points.
  The higher the achieved score, the higher is the RLS disease severity. 0 points: no symptoms, 1-10 points: mild symptoms, 11-20 points: moderate symptoms, 21-30 points: severe symptoms, 31-40 points: extreme symptoms
Time domain analysis of heart rate variability | Two days
  The standard deviation of the RR intervals (SDNN) and the root mean square of successive differences (RMSSD) in milliseconds.
Spectral analysis of heart rate variability | Two days
  The normalized high frequency component of the RR intervals (HF-HRV) is expressed as a percentage.
Spontaneous baroreceptor sensitivity | Two days
  The average baroreceptor sensitivity in ms/mmHg.

SECONDARY OUTCOMES:
Serum cytokine concentrations | Two days
  Interleukin-6, interleukin-8, interleukin-1ß and tumor necrosis factor alpha in pg/ml.
Hospital Anxiety and Depression scale | Two days
  This questionnaire has 14 items that evaluate depression and anxiety symptoms. Each item has four possible responses and is scored in a range from zero to three with higher scores representing more symptoms.
Median nerve stimulation | Two days
  Electrical nerve stimulation of the median nerve to assess its strength-duration time constant (SDTC) or chronaxie in milliseconds. The SDTC is a measure of axonal excitability and provides indirect information about the functionality of sodium ion channels.
Sudoscan | Two days
  Measurement of electrochemical skin conductance
Brief Pain Inventory | Two days
  This questionnaire assesses pain severity, location of pain, and impact on daily functions in the past 24 hours. Pain severity is scored on a numeric scale from zero to ten, with zero being no pain and ten being the worst possible pain.
Short Form 12 (SF-12) | Two days
  This questionnaire assesses the quality of life using 12 items. Each item is scaled on a range between zero and a maximum of six. Weighted sums are calculated and transformed into a population-standardized score ranging between zero and 100. The higher the score, the better is the respective life quality compared to the average population.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, Prof., Principal Investigator — University of Göttingen; Elisabeth Veiz, M.Sc., Principal Investigator — University of Göttingen; Christoph Herrmann-Lingen, Prof., Principal Investigator — University of Göttingen
Locations (1):
- University Medical Center, Göttingen, Germany

REFERENCES:
- [Derived] Veiz E, Kieslich SK, Czesnik D, Herrmann-Lingen C, Meyer T, Staab J. Increased Concentrations of Circulating Interleukins following Non-Invasive Vagus Nerve Stimulation: Results from a Randomized, Sham-Controlled, Crossover Study in Healthy Subjects. Neuroimmunomodulation. 2022;29(4):450-459. doi: 10.1159/000524646. Epub 2022 May 16. PMID 35576915